CLINICAL TRIAL: NCT05615428
Title: FAST TRIAL 2 -Fourier-transform Infrared Spectroscopy(FTIR)Guided Surfactant Therapy - Validation Study
Brief Title: Fast Assessment of Surfactant Deficiency in Preterm Infants to Speed up Treatment - Validation Study
Acronym: FAST2
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Odense University Hospital (Other); Aalborg University Hospital (Other); Aarhus University Hospital (Other); Holbaek Sygehus (Other)
Responsible Party: Principal Investigator, Christian Heiring, Principle Investigator, Rigshospitalet, Denmark
Other Study IDs: H-22007105 Validation Study
Record Dates: First submitted 2022-11-07; First posted 2022-11-14 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2024-09

CONDITIONS: Surfactant Deficiency Syndrome Neonatal; Respiratory Distress Syndrome in Premature Infant
Keywords: surfactant replacement therapy; surfactant assay
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Gastric aspirate from newborn infants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- observational group: Inclusion criteria:
  * GA ≤29+6, inborn at a participating centre
  * Age less than 45 minutes as gastric aspirate must be sampled within 45 minutes from delivery.
  Exclusion criteria:
  * Treated with surfactant beforerandomisation and obtaining gastric aspirates
  * Diagnosis of major malformations (major congenital heart defects, congenital diaphragmatic hernia, gastroschisis/omphalocele, pulmonary abnormalities including pulmonary hypoplasia and trachea-oesophageal fistula
  * Antenatal suspicion of significant oligohydramnios and lung hypoplasia
  * Any intrauterine intervention except if done for genetic testing
  Interventions: Diagnostic Test: LS-ratio

INTERVENTIONS:
Diagnostic Test: LS-ratio — Included infants will have a gastric aspirate sampled via an NG tube at birth. This sample will be analyzed to determine the LS-ratio The LS-ratio will retrospectively be compared to RDS development and need for surfactant treatment to establish the cut-off ratio for LS-ratio with respect to surfactant treatment.

SUMMARY:
The aim is to re-validate a FTIR spectroscopy test for measuring lung maturity/Respiratory Distress Syndrome (RDS) before conducting a RCT using this test to guide surfactant treatment of preterm infants.

The test has been validated previously (NCT03235882) but needs re-validation due to continued improvement in accuracy and since the test is now developed into a Point of Care test (POC-test).

The purpose is to accurately predict RDS using Lecithin/Sphingomyelin ratio (L/S ratio determined by a rapid FTIR in a newly developed point of care test (POC-test) on fresh gastric aspirates using retrospective analysis.

The FAST 2 Validation Study is a part of the FAST 2 Trial consisting of a validation study and a subsequent randomized clinical trial, that will be registered separately on clinicaltrials.gov (NTC XXXXXXXXX)

DETAILED DESCRIPTION:
Treatment of respiratory distress syndrome (RDS) has evolved greatly over the past three decades. Major advances in treatment include antenatal steroids, early nasal continuous positive airway pressure (nCPAP) combined with early rescue surfactant replacement strategies such as Intubation Surfactant Extubation (INSURE) and Less Invasive Surfactant Administration (LISA), together with use of lung protective ventilation and overall reduced use of mechanical ventilation. However, RDS and bronchopulmonary dysplasia (BPD) are still major causes of mortality and morbidity in premature infants. To improve the outcome, very early treatment with surfactant is necessary. However, only about half of infants with a gestational age (GA) below 30 weeks need surfactant treatment and prophylactic surfactant treatment increases the combined mortality and incidence of BPD contrary to selective rescue surfactant treatment. Therefore, there is a need for a rapid test to guide early targeted surfactant treatment.

We have recently developed a new test of lung maturity based on measuring the lecithin sphingomyelin ratio (L/S) in fresh gastric aspirates (GAS) from newborn preterm infants using mid-red Fourier Transform Infrared spectroscopy (FTIR). The sphingomyelin concentration in amniotic fluid and accordingly in GAS is relatively constant during the pregnancy, whereas the lecithin (or dipalmitoylphosphatidylcholine (DPPC), the lung surfactant phospholipid with the highest surface activity) concentration increases with the lung maturation.

We have demonstrated in clinical observational trials that our laboratory based L/S-test predicts development of RDS when measured immediately at delivery (FAST 1 Trial).

The L/S-test has now been developed into an easy-to-use Point of Care (POC) test for bedside use that expresses the L/S ratio in approximately 10 minutes. We believe this new POC test can be used to guide surfactant therapy, enabling very early rescue treatment, potentially even before symptoms occur.

To obtain evidence-based knowledge on harms and benefit of surfactant therapy guided by the L/S test, a randomized clinical trial with relevant clinical short-and long-term outcomes needs to be performed, which is why the FAST 2 Trial has been designed.

During design and development of the FAST 2 Trial protocol extensive engineering work has been conducted towards building a fully automated L/S POC Device (AIMI 1.0/2.0) from the prototypes in the first L/S studies (including FAST 1 Trial).

During this process the accuracy of the L/S algorithm has been improved through machine learning and use of artificial intelligence. Consequently, the previously defined cut-off ratio from the FAST 1 Trial needs to be re-validated using the L/S POC Device in a new population of preterm infants.

The FAST 2 Trial therefore consists of two individual studies starting with the FAST 2 Validation Study which will followed by the FAST 2 Randomized Clinical Trial (FAST 2 RCT) once completed. The FAST 2 RCT will be registered at clinicaltrials.gov separately.

The objective of FAST 2 Validation study is:

In preterm infants with gestational age at birth of ≤ 29+6 weeks less than 45 minutes of age who have not received surfactant prior to the measurenent, we aim to:

• measure L/S-ratio in fresh GAS using the AIMI 1.0/2.0 L/S POC Device

and compare the L/S-ratio by: • the need for surfactant treatment

with the aim to:

• validate the previously defined optimal cut-off L/S-ratio for surfactant treatment and to determine if the cut-off L/S ratio needs to be adjusted before starting FAST 2 RCT

ELIGIBILITY:
Inclusion Criteria:

GA ≤29+6, inborn at a participating centre Age less than 45 minutes as gastric aspirate must be sampled within 45 minutes from delivery.

Exclusion criteria:

Treated with surfactant beforerandomisation and obtaining gastric aspirates

Diagnosis of major malformations (major congenital heart defects, congenital diaphragmatic hernia, gastroschisis/omphalocele, pulmonary abnormalities including pulmonary hypoplasia and trachea-oesophageal fistula

Antenatal suspicion of significant oligohydramnios and lung hypoplasia

Any intrauterine intervention except if done for genetic testing

Max Age: 45 Minutes | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm newborn babies that have gastric secretions sampled before 45 minutes of age.
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2023-02-16 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
LS-ratio cut-off | 5 days
  The primary objective is to measure the L/S-ratio in fresh GAS using the AIMI 1.0/2.0 L/S POC Device and compare the L/S-ratio with the need for surfactant treatment aiming to validate the previously defined cut-off L/S-ratio for surfactant treatment and to determine if the cut-off L/S ratio needs adjustment before starting FAST 2 RCT

CONTACTS AND LOCATIONS:
Overall Officials: Christian Heiring, Principal Investigator — Rigshospitalet, Denmark
Locations (3):
- Denmark (3):
  - Aalborg University Hospital, Aalborg
  - Aarhus University Hospital, Aarhus
  - Odense University Hospital, Odense

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol